CLINICAL TRIAL: NCT00087698
Title: A Multicenter Phase II Trial of Neo-Adjuvant Pemetrexed (Alimta) Plus Cisplatin Followed by Surgery and Radiation for Pleural Mesothelioma
Brief Title: Phase II Trial of Neo-Adjuvant Pemetrexed Plus Cisplatin Followed by Surgery and Radiation for Pleural Mesothelioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7216; H3E-US-JMGA; NCT00072397 (obsolete NCT alias)
Record Dates: First submitted 2004-07-12; First posted 2004-07-16 (Estimated); Results first posted 2009-03-17 (Estimated); Last update posted 2009-05-12 (Estimated); Status verified 2009-05

CONDITIONS: Pleural Neoplasms
MeSH Terms: conditions — Pleural Neoplasms | interventions — Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): chemotherapy, surgery then chest radiation x 54 gray (Gy)
  Interventions: Drug: pemetrexed; Drug: cisplatin

INTERVENTIONS:
Drug: pemetrexed — 500 mg/m2, intravenous (IV), every 21 days x 4 cycles
  Other Names: LY231514; Alimta
Drug: cisplatin — 75 mg/m2, intravenous (IV), every 21 days x 4 cycles

SUMMARY:
This study aims to determine how successful the chemotherapy regimen of Pemetrexed plus cisplatin before surgery is at killing all the tumor so that none is left at the time of surgery. Following surgery, all eligible patients will receive radiation to the chest. How patients respond, whether the cancer returns and if so, where, will also be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be clinically staged using AJCC/UICC TNM staging criteria. Eligible stages:

  1. Patients must be M0
  2. Patients with T1, T2, and T3 disease (without cardiac involvement) are eligible (T status can be established clinically and radiologically or at exploratory thoracotomy without surgical resection
  3. Patients with N0, N1,or N2 disease are eligible
* Performance status of 0 to 1 on the ECOG performance status schedule.
* No prior systemic chemotherapy and no prior intracavitary cytotoxic drugs or immunomodulators, unless given for the purpose of chemical pleurodesis
* No previous radiation therapy
* Estimated life expectancy of at least 12 weeks

Exclusion Criteria:

Patients will be excluded if they meet ANY of the following criteria:

* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry
* Have previously completed or withdrawn from this study or any other study investigating pemetrexed
* Pregnancy or breast-feeding
* Serious concomitant systemic disorders (i.e. active infection) that, in the opinion of the investigator, would compromise the safety of the patient or compromise the patient's ability to complete the study
* Second active primary malignancy (except in situ carcinoma of the cervix, adequately treated non-melanomatous carcinoma of the skin, low grade (Gleason score less than or equal to 6), localized adenocarcinoma of the prostate or other malignancy treated at least 2 years previously with no evidence of recurrence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2003-09; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- United States (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Francisco, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boston, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Detroit, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas

REFERENCES:
- [Derived] Federico R, Adolfo F, Giuseppe M, Lorenzo S, Martino DT, Anna C, Adriano P, Gino C, Francesca R, Matteo C, Gbenga K, Paolo M, Francesco F. Phase II trial of neoadjuvant pemetrexed plus cisplatin followed by surgery and radiation in the treatment of pleural mesothelioma. BMC Cancer. 2013 Jan 16;13:22. doi: 10.1186/1471-2407-13-22. PMID 23324131
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Pemetrexed: pemetrexed: 500 mg/m2, intravenous, every 21 days x 4 cycles cisplatin: 75 mg/m2, intravenous, every 21 days x 4 cycles chemotherapy, surgery then chest radiation x 54 gray (Gy)
Period: Overall Study
Arm/Group | Pemetrexed
Started | 77
Completed | 41
Not Completed | 36
Not completed — Lack of Efficacy, Progressive Disease | 14
Not completed — Death from Other Causes | 3
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 4
Not completed — Lack of Efficacy, Physician Perception | 3
Not completed — Protocol Entry Criteria Not Met | 2
Not completed — Clinical Relapse | 1
Not completed — Death from Study Disease | 2
Not completed — Death from Study Drug Toxicity | 2
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pemetrexed
Number analyzed (Participants) | 77
Age Continuous [Mean (Standard Deviation); unit: years] | 61.1 (9.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 56
Region of Enrollment [Number; unit: participants]
  United States | 77
Disease Stage at Time of Study Entry [Number; unit: participants]
  Stage IA | 3
  Stage IB | 3
  Stage II | 33
  Stage III | 35
  Stage IV | 1
  Unknown/Not Available | 2
Eastern Cooperative Oncology Group Performance Status [Number; unit: participants]
  0 - Fully active and asymptomatic | 28
  1 - Ambulatory with symptoms | 47
  2 - In bed < 50% of time | 2
Initial Pathological Diagnosis [Number; unit: participants]
  Epithelial Mesothelioma | 62
  Mixed Cell Mesothelioma | 2
  Sarcomatoid Mesothelioma | 1
  Other | 12
Race/Ethnicity [Number; unit: participants]
  Caucasian | 71
  African | 1
  East/Southeast Asian | 1
  Western Asian | 2
  Hispanic | 2
Time from Initial Pathological Diagnosis to Enrollment [Mean (Standard Deviation); unit: months] | 2.19 (2.909)

OUTCOME MEASURES:

1. Primary Outcome: Pathological Complete Response
Description: Number of participants with results of pathological review that indicated a complete response. Pathological complete response should be evaluated at the time of surgery (Extrapleural Pneumonectomy [EPP]).
  Resected tissue or pleural fluid should be sent for pathological and histological evaluation.
Time Frame: Surgery (at least 3 weeks post last dose of chemotherapy, up to a maximum interval of 8 weeks)
Population: All participants who had undergone surgery.
Measure: Number; unit: participants
Arm/Group | Pemetrexed
Number analyzed (Participants) | 57
participants | 3

2. Secondary Outcome: The 1 and 2 Year Disease-Free Survival Rate (Percentage)
Description: Kaplan-Meier estimates of the percentage of participants still alive at 1-year and 2-years, based upon the total number of participants who had surgery.
Time Frame: 1 year and 2 years
Population: All participants who had undergone surgery.
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed
Number analyzed (Participants) | 57
percentage of participants
  1-Year Disease-Free Rate | 61.40 [47.53 to 72.63]
  2-Year Disease-Free Rate | 33.24 [21.45 to 45.47]

3. Secondary Outcome: Overall Tumor Response
Description: The frequency of best overall tumor response summarized by response category. The best (unconfirmed) response recorded from the start of chemotherapy treatment until disease progression/recurrence, start of any further anti-tumor therapy, or time of surgery whichever comes first.
Time Frame: baseline to measured progressive disease
Population: Intention to Treat analysis. All enrolled participants who were eligible for the treatment, whether or not they received the study drug.
Measure: Number; unit: participants
Arm/Group | Pemetrexed
Number analyzed (Participants) | 77
participants
  Complete Response | 1
  Partial Response | 24
  Stable Disease | 36
  Progressive Disease | 5
  Unknown/Unavailable | 11

4. Secondary Outcome: Time to Treatment Failure
Description: Time to relapse (treatment failure) is measured in months and calculated as (Date of first surgery - Date of first relapse after surgery + 1)/(365.25/12). Time to relapse will be censored at the date of the last visit or start date of further anti-tumor therapy or intervention, whichever comes first.
Time Frame: baseline to stopping treatment
Population: All participants who had undergone surgery.
Measure: Mean (Full Range); unit: months
Arm/Group | Pemetrexed
Number analyzed (Participants) | 57
months | 18.30 [1.71 to 41.89]

5. Secondary Outcome: Time to Progressive Disease
Description: Number of months between the first dose date and the date of first disease progression or death as a result of any cause, whichever comes first.
Time Frame: baseline to measured progressive disease
Population: All participants who had undergone surgery.
Measure: Mean (Full Range); unit: months
Arm/Group | Pemetrexed
Number analyzed (Participants) | 57
months | 14.98 [2.56 to 46.00]

6. Secondary Outcome: Overall Survival Time
Description: Number of months between the first dose date and the date of death as a result of any cause. Overall survival time calculated as (Date of death - First dose date + 1)/(365.25/12).
Time Frame: baseline to date of death from any cause
Population: All participants who had undergone surgery.
Measure: Mean (Full Range); unit: months
Arm/Group | Pemetrexed
Number analyzed (Participants) | 57
months | 21.85 [3.25 to 46.00]

ADVERSE EVENTS:
Groups:
- Pemetrexed: pemetrexed: 500 mg/m2, intravenous (IV), every 21 days x 4 cycles cisplatin: 75 mg/m2, intravenous (IV), every 21 days x 4 cycles chemotherapy, surgery then chest radiation x 54 Gy
Arm/Group | Pemetrexed
Serious Adverse Events (participants affected / at risk) | 15
Other Adverse Events (participants affected / at risk) | 77
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Pemetrexed
Febrile neutropenia (Blood and lymphatic system disorders) | 2/77 (2)
Atrial fibrillation (Cardiac disorders) | 1/77 (1)
Sinus bradycardia (Cardiac disorders) | 1/77 (1)
Vomiting (Gastrointestinal disorders) | 2/77 (2)
Chest pain (General disorders) | 1/77 (3)
Death (General disorders) | 1/77 (1)
Infection (Infections and infestations) | 1/77 (1)
Pneumonia (Infections and infestations) | 4/77 (5)
Blood creatinine increased (Investigations) | 2/77 (2)
Anorexia (Metabolism and nutrition disorders) | 1/77 (1)
Dehydration (Metabolism and nutrition disorders) | 1/77 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1/77 (1)
Renal failure (Renal and urinary disorders) | 1/77 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1/77 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2/77 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2/77 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1/77 (1)
Deep vein thrombosis (Vascular disorders) | 1/77 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Pemetrexed
Anaemia (Blood and lymphatic system disorders) | 17/77 (22)
Leukopenia (Blood and lymphatic system disorders) | 5/77 (8)
Neutropenia (Blood and lymphatic system disorders) | 8/77 (10)
Tachycardia (Cardiac disorders) | 7/77 (7)
Tinnitus (Ear and labyrinth disorders) | 12/77 (13)
Lacrimation increased (Eye disorders) | 5/77 (5)
Vision blurred (Eye disorders) | 5/77 (6)
Abdominal distention (Gastrointestinal disorders) | 4/77 (6)
Abdominal pain (Gastrointestinal disorders) | 5/77 (6)
Constipation (Gastrointestinal disorders) | 45/77 (62)
Diarrhoea (Gastrointestinal disorders) | 20/77 (21)
Dyspepsia (Gastrointestinal disorders) | 8/77 (9)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4/77 (4)
Nausea (Gastrointestinal disorders) | 57/77 (87)
Stomatitis (Gastrointestinal disorders) | 15/77 (15)
Vomiting (Gastrointestinal disorders) | 34/77 (47)
Chest discomfort (General disorders) | 7/77 (8)
Chest pain (General disorders) | 9/77 (10)
Chills (General disorders) | 5/77 (5)
Fatigue (General disorders) | 51/77 (79)
Oedema peripheral (General disorders) | 9/77 (12)
Pain (General disorders) | 5/77 (5)
Pyrexia (General disorders) | 10/77 (12)
Drug hypersensitivity (Immune system disorders) | 6/77 (8)
Blood creatinine increased (Investigations) | 6/77 (8)
Breath sounds abnormal (Investigations) | 8/77 (8)
Haemoglobin decreased (Investigations) | 4/77 (4)
Weight decreased (Investigations) | 4/77 (5)
White blood cell count decreased (Investigations) | 4/77 (4)
Anorexia (Metabolism and nutrition disorders) | 22/77 (25)
Decreased appetite (Metabolism and nutrition disorders) | 6/77 (6)
Dehydration (Metabolism and nutrition disorders) | 4/77 (4)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 4/77 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 6/77 (7)
Hypomagnesaemia (Metabolism and nutrition disorders) | 6/77 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10/77 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 5/77 (6)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4/77 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 5/77 (5)
Dizziness (Nervous system disorders) | 7/77 (7)
Dysgeusia (Nervous system disorders) | 16/77 (16)
Headache (Nervous system disorders) | 10/77 (13)
Neuropathy (Nervous system disorders) | 5/77 (6)
Parosmia (Nervous system disorders) | 4/77 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 5/77 (5)
Anxiety (Psychiatric disorders) | 8/77 (8)
Insomnia (Psychiatric disorders) | 10/77 (10)
Pollakiuria (Renal and urinary disorders) | 4/77 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 18/77 (19)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12/77 (12)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5/77 (5)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 6/77 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 8/77 (8)
Night sweats (Skin and subcutaneous tissue disorders) | 6/77 (6)
Rash (Skin and subcutaneous tissue disorders) | 18/77 (24)
Flushing (Vascular disorders) | 5/77 (5)
Hypertension (Vascular disorders) | 6/77 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days